CLINICAL TRIAL: NCT01614067
Title: Delayed Start to Ovarian Stimulation Improves Oocyte Maturation and Quality: A Randomized Trial
Brief Title: Delayed Start to Ovarian Stimulation
Acronym: DOS/DOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment resulted in withdraw of funding
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSF 11-07259
Record Dates: First submitted 2012-05-02; First posted 2012-06-07 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Diminished Ovarian Reserve; Infertility; In Vitro Fertilization
Keywords: DOR; Infertility; IVF; ART; GnRHa; GnRH Antagonist Protocol; Ganirelix
MeSH Terms: conditions — Infertility | interventions — ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Delayed Start (Experimental): Study subjects will receive 7 days of pre-treatment with a GnRH antagonist (Delayed Start) before standard ovarian stimulation with FSH/LH.
  Interventions: Drug: Ganirelix acetate
- Conventional Start (Active Comparator): Ovarian stimulation with standard antagonist protocols (no delay).
  Interventions: Drug: Ganirelix acetate

INTERVENTIONS:
Drug: Ganirelix acetate — Subjects will receive 7 days of pre-treatment with the GnRH antagonist
  Other Names: Ganirelix

SUMMARY:
In couples with infertility secondary to Diminished Ovarian Reserve, the investigators hypothesize that a delayed start (7 day) to ovarian stimulation with an GnRH antagonist (Ganirelix) will improve oocyte maturation and quality, and improve pregnancy outcomes.

DETAILED DESCRIPTION:
Over the past two decades, the success rate of assisted reproductive technology (ART) has dramatically increased. This increase is attributed to improvements in embryo culture, laboratory conditions, and optimization of ovarian stimulation protocols. Over the past years, there has been more interest in altering the ovarian stimulation protocol to improve outcomes. For example, recently our group found that a modification of ovulation trigger toward a more physiologic process improves oocyte quality and pregnancy outcomes. Others have suggested minimal stimulation improves in vitro fertilization (IVF) outcomes. The investigators propose to further investigate modifying the ovarian stimulation for women who have "decreased" ovarian reserve. The investigators propose that a delayed start to ovarian stimulation will improve oocyte maturation and quality and pregnancy outcomes. No published studies to date have evaluated if a delayed start to ovarian stimulation improves pregnancy outcomes. However, the investigators hypothesize that the use an antagonist for a delayed start of stimulation will work by one of two mechanisms:

I. The partial suppression of FSH will allow for further recruitment of early antral follicles.

II. The partial suppression of FSH will allow for further FSH responsiveness in existing follicles to synchronize the primary cohort, thereby increasing the total number of follicles.

ELIGIBILITY:
Inclusion Criteria:

* Antral Follicle Count (AFC) less than or equal to 4 as measured by transvaginal ultrasound (TVUS), or
* Cancellation of a prior IVF cycle due to poor ovarian response.
* Patients will receive an antagonist stimulation protocol for IVF, or IVF with Intracytoplasmic Sperm Injection (ICSI).

Exclusion Criteria:

* Severe male factor infertility requiring surgical intervention to obtain sperm
* Major uterine abnormality,
* Preimplantation genetic diagnostic (PGD) testing,
* Planned cycles without embryo transfer (for example, freeze-all, donor, or surrogate cycles).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, MD, Principal Investigator — UCSF Center for Reproductive Health and Fertility Preservation
Locations (1):
- UCSF Center for Reproductive Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blockeel C, Riva A, De Vos M, Haentjens P, Devroey P. Administration of a gonadotropin-releasing hormone antagonist during the 3 days before the initiation of the in vitro fertilization/intracytoplasmic sperm injection treatment cycle: impact on ovarian stimulation. A pilot study. Fertil Steril. 2011 Apr;95(5):1714-9.e1-2. doi: 10.1016/j.fertnstert.2011.01.028. PMID 21300334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With a goal of enrolling a total of 114 subjects, 330 potential candidates were screened for eligibility. 300 candidates were either not eligible or declined participation. 30 subjects were found eligible to participate and enrolled in the study.
Period: Overall Study
Arm/Group | Delayed Start | Conventional Start
Started (Arm randomization assignment prior to starting clinical treatment cycle) | 15 | 15
Completed | 0 | 0
Not Completed | 15 | 15
Not completed — Pregnancy | 1 | 0
Not completed — Physician Decision | 6 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study terminated early by sponsor and was unable to collect data | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Start | Conventional Start | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants] — Female patients ages 18 years and older who were seeking IVF treatment.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 15 | 30
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Fertilization Proportions
Description: Developmental competence (fertilization of oocytes) through standard in vitro fertilization (estimated time frame to be between 8-24 hours following IVF). This percentage will be calculated as the number of fertilized eggs ( 2PN stage) per total number of eggs collected from the egg retrieval.
Time Frame: 8 to 24 hours after in vitro fertilization, oocytes will be checked for fertilization
Population: The study was terminated early and no data were collected for this outcome measure
Arm/Group | Delayed Start | Conventional Start
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Oocytes Retrieved
Description: The egg retrieval procedure will be performed 36 hours after the ovulation trigger. The procedure is estimated to take up to 1 hour at study visit as part of routine care. The number of retrieved eggs will be counted
Time Frame: up to 1 hour after oocytes retrieved
Population: The study was terminated early and no data were collected for this outcome measure
Arm/Group | Delayed Start | Conventional Start
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Embryo Quality
Description: Embryo quality will be assessed by the embryologist on days 2 or 3 (Cleavage stage) following IVF using standard embryo grading criteria. Embryos grading is based on three criteria: the number of blastomere cells present in the embryo, the degree of observed cell fragmentation and the degree of observed symmetry of the cells.
Time Frame: One hour on day 2 or 3 (following IVF procedure)
Population: The study was terminated early and no data were collected for this outcome measure
Arm/Group | Delayed Start | Conventional Start
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pregnancy Rates
Description: Beta HCG levels will be assessed at 2 weeks and 3 weeks after embryo transfer. A positive pregnancy is defined as two positive beta HCG levels (a value > 5 mIU/ml ) observed over the time frame.
Time Frame: 2 to 3 weeks following embryo transfer
Population: The study was terminated early and no data were collected for this outcome measure
Arm/Group | Delayed Start | Conventional Start
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Stages of Oocyte Nuclear Maturation
Description: Quality of oocytes will be assessed for developmental stages (Germinal Vesicles, Meiosis I, or Meiosis II)
Time Frame: average of 1 to 2 hours on the Day of Retrieval
Population: The study was terminated early and no data were collected for this outcome measure
Arm/Group | Delayed Start | Conventional Start
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Mature Follicles
Description: Maturation of follicles will be assessed by measuring the size of follicles (mature > 13mm) prior to (or at the time of) oocytes retrieval.
Time Frame: up to 1 hour (during the Transvaginal Ultrasound before Retrieval of Oocytes)
Population: The study was terminated early and no data were collected for this outcome measure
Arm/Group | Delayed Start | Conventional Start
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Oocyte Recovery Rate
Description: The number of oocytes recovered at the time of oocyte retrieval following ovarian stimulation.
Time Frame: up to 1 hours after oocyte retrieval
Population: The study was terminated early and no data were collected for this outcome measure
Arm/Group | Delayed Start | Conventional Start
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Delayed Start | Conventional Start
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No